CLINICAL TRIAL: NCT00752830
Title: A Phase I, Open, Randomized, Single-Dose, Two-Treatment (Fed Versus Fasting), Two-Period Cross-Over Single-Centre Study to Evaluate the Effect of Food on the Pharmacokinetics of AZD0328 Following Oral Administration (Capsule) in Healthy Male Subjects
Brief Title: To Evaluate the Effect of Food on the Pharmacokinetics (PK) of AZD0328
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Didier Meulien, MD, Medical Science Director, Emerging AD & Cognition, AstraZeneca R&D, Södertälje, Sweden
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D0190C00009; EUdract NO 2008-003691-22
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: AZD0328; Food Effect
MeSH Terms: interventions — spiro(1-azabicyclo(2.2.2)octane-3,2'(3H)-furo(2,3-b)pyridine)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD0328 administration during fasting condition
  Interventions: Drug: AZD0328
- 2 (Experimental): AZD0328 administration after food intake
  Interventions: Drug: AZD0328

INTERVENTIONS:
Drug: AZD0328 — Oral capsule, single dose

SUMMARY:
The purpose of the study is to evaluate the effect of food on the pharmacokinetics of AZD0328 in healthy male volunteers. AZD0328 will be administered as a single oral dose (capsule) during two treatment periods, after food intake or during fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Caucasian subjects.
* Clinically normal physical findings, laboratory values, vital signs and resting ECG as judged by the investigator.
* Signed informed consent form

Exclusion Criteria:

* History of clinically significant cardio or cerebrovascular, pulmonary, renal, hepatic, neurological, mental or gastrointestinal disorder (including dyspepsia or GERD) or any other major disorder that may interfere with the study.
* Intake of another investigational drug or participation in another study which may interfere with the objectives of the study, within 12 weeks before the administration of the investigational product.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
PK variables | Several PK samples during the study days

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, laboratory measurements and paper ECGs) | During the whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Didier Meulien, MD, Study Director — AstraZeneca R&D Södertälje, Sweden; Gabriella Samuelsson Palmgren, MD, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, AstraZeneca R&D Lund,Sweden
Locations (1):
- Research Site, Lund, Sweden